CLINICAL TRIAL: NCT02589886
Title: Self-Help and Education on the Internet for Functional Motor Disorders, a Randomised Controlled Trial (SHIFT)
Brief Title: Self-help and Education on the Internet for Functional Motor Disorders
Acronym: SHIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Marina de Koning-Tijssen, Prof. Dr. de Koning-Tijssen, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: METc/2015/141
Record Dates: First submitted 2015-10-02; First posted 2015-10-28 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Functional Motor Disorder
Keywords: Self-help; Education; e-Health
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Active Comparator): This arm will receive the education and self-help internet intervention added to usual care
  Interventions: Other: Education and self-help internet intervention
- control (No Intervention): This arm will receive usual care only

INTERVENTIONS:
Other: Education and self-help internet intervention — The intervention is a newly developed website which consists of information about the mechanism and treatment of functional motor disorders. Furthermore self-help elements like exercises to perform at home and rehabilitation advice are added. The intervention is unguided.
  Arms: intervention

SUMMARY:
A randomised trial to the effect of a newly developed education and self help intervention for patients with a functional motor disorder on general health, quality of life, illness perception, symptom severity and other secondary outcome measures.

DETAILED DESCRIPTION:
Patients will be referred to the study from all neurology centers in the Netherlands that are found willing to participate. After informed consent is acquired, patients will be randomised into one of these two groups: usual care only or the education and self help intervention added to usual care. At baseline, after 3 months and after 6 months patients will fill out questionnaires at home online or on paper.

Patients will not be blinded for the intervention. The researcher is blinded during analysis of the data. During the study contact between the researcher and the participants will be restricted to research related topics. All contact between participants and the researcher will be documented.

To increase generalisability and applicability in clinical practice after the trial the investigators have chosen to add the intervention to usual care and to keep exclusion criteria to a minimum.

Our education and self help internet intervention is an especially designed website with an educational approach. The content of the intervention is written by a team of international experts and consists of education about the mechanism of functional motor disorders and it's treatment and of self help advice and exercises. During the trial the website will only be accessible with a log-in. The education and self help internet intervention is self-explanatory and unguided.

The medical ethical committee of the University Medical Center Groningen has taken our research under review and has decided this study does not fall under the scope of the Medical Research Involving Human Subjects Act (WMO-Wet Mensgebonden Onderzoek).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of functional motor symptom from a neurologist
* The motor symptom(s) cause(s) distress or impairment in social, occupational or other important areas of functioning.
* Able to read Dutch
* Access to a computer with internet connection on a regular basis

Exclusion Criteria:

* Incapacitated (Not able to provide informed consent)
* Accidental finding of a motor symptom in a patient with other (functional) complaints.
* Known existing visitor of the (previously available, but currently offline) translated version of a website by Dr. Jon Stone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Subjective general health Status on the Clinical Global Improvement scale | 3 months
  CGI, self-rated, 7-point scale of general health status
Subjective general health Status on the Clinical Global Improvement scale | 6 months
  CGI self-rated, 7-point scale of general health status

SECONDARY OUTCOMES:
Quality of life on domains of RAND-36 | 3 months
  extra question added to RAND-36 from WHOQuality Of Life scale
Quality of life on domains of RAND-36 | 6 months
  extra question added to RAND-36 from WHO-Quality Of Life scale
Illness beliefs on the Illness Perception Questionnaire | 3 months
  Questions from the Illness Perception Questionnaire and newly devised questions about beliefs and understanding of functional motor disorders
Illness beliefs on the Illness Perception Questionnaire | 6 months
  Questions from the Illness Perception Questionnaire and newly devised questions about beliefs and understanding of functional motor disorders
Referral and other treatments on a questionnaire about referral and other treatments | 6 months
  Questions about future and past referrals to treatment
Symptom severity on the change in presenting symptoms scale | 3 months
Symptom severity on the change in presenting symptoms scale | 6 months
Work and social adjustment | 6 months
  Work and Social Adjustment scale
Cost-effectivity in QALY's calculated by using the PCQ, MCQ and EQ5D | 6 months
  Analysis using: Patient Costs Questionnaire, Medical Costs Questionnaire, and EQ5D
Patient satisfaction with general care and the study intervention | 3 months
  Questions on satisfaction with general care and with the education and selfhelp intervention in particular
Patient satisfaction with general care and the study intervention | 6 months
  Questions on satisfaction with general care and with the education and selfhelp intervention in particular
Psychiatric outcome on the Patient Health Questionnaire | 6 months
Fatigue on CIS-fatigue scale | 6 months

OTHER OUTCOMES:
Adverse events | 6 months
  Death and hospitalization during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Marina Tijssen, MD, PhD, Principal Investigator — University Medical Center Groningen, University of Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sharpe M, Walker J, Williams C, Stone J, Cavanagh J, Murray G, Butcher I, Duncan R, Smith S, Carson A. Guided self-help for functional (psychogenic) symptoms: a randomized controlled efficacy trial. Neurology. 2011 Aug 9;77(6):564-72. doi: 10.1212/WNL.0b013e318228c0c7. Epub 2011 Jul 27. PMID 21795652
- [Background] Lehn A, Gelauff J, Hoeritzauer I, Ludwig L, McWhirter L, Williams S, Gardiner P, Carson A, Stone J. Functional neurological disorders: mechanisms and treatment. J Neurol. 2016 Mar;263(3):611-20. doi: 10.1007/s00415-015-7893-2. Epub 2015 Sep 26. PMID 26410744
- [Background] Stone J, Carson A. Functional neurologic disorders. Continuum (Minneap Minn). 2015 Jun;21(3 Behavioral Neurology and Neuropsychiatry):818-37. doi: 10.1212/01.CON.0000466669.02477.45. PMID 26039857
- [Background] Gelauff JM, Dreissen YE, Tijssen MA, Stone J. Treatment of functional motor disorders. Curr Treat Options Neurol. 2014 Apr;16(4):286. doi: 10.1007/s11940-014-0286-5. PMID 24566832
- [Derived] Gelauff JM, Rosmalen JGM, Carson A, Dijk JM, Ekkel M, Nielsen G, Stone J, Tijssen MAJ. Internet-based self-help randomized trial for motor functional neurologic disorder (SHIFT). Neurology. 2020 Sep 29;95(13):e1883-e1896. doi: 10.1212/WNL.0000000000010381. Epub 2020 Jul 20. PMID 32690783